CLINICAL TRIAL: NCT02588924
Title: Study on the Relationship Between Environmental and Occupational Exposure to Metals and Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, PAOLA PEDATA, Universitary researcher of Second University of Naples, University of Campania Luigi Vanvitelli
Other Study IDs: 961
Record Dates: First submitted 2015-09-28; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Parkinson Disease, Secondary
Keywords: Parkinson Disease; ENVIRONMENTAL AND OCCUPATIONAL EXPOSURE TO METALS
MeSH Terms: conditions — Parkinson Disease, Secondary; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Second University of Naples: the present research project is aimed at measuring out the concentrations of copper, iron and manganese in biological fluids (blood, serum) of patients with Parkinson's disease and of subjects of the control group and assess possible correlations between changes in the content of metals and the pathology.
  Interventions: Other: Second University of Naples
- Neuromed IRCCS: the present research project is aimed at measuring out the concentrations of copper, iron and manganese in biological fluids (blood, serum) of patients with Parkinson's disease and of subjects of the control group and assess possible correlations between changes in the content of metals and the pathology.
  Interventions: Other: Neuromed IRCCS

INTERVENTIONS:
Other: Second University of Naples — enrollment of patients with Parkinson's disease; collection of blood samples; measuring out the concentrations of copper, iron and manganese in biological fluids (blood, serum) of patients with Parkinson's disease and of subjects of the control group and assess possible correlations between changes in the content of metals and the pathology.
  Groups: Second University of Naples
Other: Neuromed IRCCS — enrollment of patients with Parkinson's disease; collection of blood samples;
  Groups: Neuromed IRCCS

SUMMARY:
The Department of Experimental Medicine - Section of Hygiene, Occupational Medicine, Forensic Medicine of the Second University of Naples, the Section of Neurology of the Second University of Naples and the Mediterranean Neurological Institute NEUROMED, IRCCS are involved in the realization of a research project aimed at studying the correlation between environmental and occupational exposure to metals (copper, iron and manganese) and Parkinson disease in order to increase the knowledge of these possible risk factors and highlight an eventual predictive-diagnostic meaning of possible discrepancies in the content of these elements; secondly the collected data could be used for assessing the association (odd ratio-OR) between pathologies and different risk factors (for example smoking habits, professional exposure and so on).

DETAILED DESCRIPTION:
During the selection of the sample it is essential to consider all the variables that could provoke an alteration in the levels of the indicators examined in the biological fluids investigated.

The adoption of strict criteria for inclusion and exclusion, which differ from metal to metal, is therefore necessary to establish the presence / absence of possible confounding factors that could affect the analysis or interpretation of the data.

It is to be noted also that the number of required participants in a study of MB must be sufficiently large to allow an adequate statistical analysis: the more limited the group of subjects included in the study is, the broader the variability of the data due to inter-individual and methodological differences.

In light of this, some variables, such as age and sex, will be firstly neglected and other potential confounding factors will be considered such as, for example, smoking habits.

Based on the purpose of the research project, the following criteria for exclusion will be considered:

* diseases that may interfere with toxicokinetics of the analyzed metals;
* pharmacological therapy;
* habit-forming additives consumption (excessive alcohol consumption);
* altered physiological states (pregnancy, strenuous physical exercise, recent meal, stress, psychological disorders);

On the contrary, the basic criteria for inclusion in the study are:

* age: subjects of working age, between 18 and 65 years;
* diagnosis of Parkinson's disease (using the criteria of the "London Brain Bank")

Regarding the criteria of partition or stratification of the subjects, the type and number of the possible partitions are conditioned by the sample size; indeed it is essential to ensure a sufficient number of cases (and if possible a similar number of cases) in the various layers to have correct statistical results. It was recommended that the minimum number of subjects per layer must be equal to 80.

In order to collect all the necessary information for the inclusion of subjects in the study and the subsequent stratification of the data, an anonymous questionnaire was realized and administered to each recruited subject.

The questionnaire deals with the environment and the lifestyle and work habits of every participant and it consists of multiple choice questions and free response questions and is divided into macro areas: identification data for data processing; place of residence; professional activity; extraprofessional activities; eating habits; habit-forming additives consumption; medical history.

Each question will be transformed into a "continue" or "categorical" variable in order to be able to build and constantly update a database summarizing the collected data and allowing the statistical analysis of the results.

Each subject enrolled will be also asked to sign a consent form, which states that he or she voluntarily take part to the study, after being informed about the purpose of the study and the analysis of both biological samples and personal data.

The guarantee of anonymity for people recruited for this study is provided by an anonymous questionnaire which do not contain personal data, which are collected only in the consent form, separately from the questionnaire.

ELIGIBILITY:
EXCLUSION CRITERIA:

* diseases that may interfere with toxicokinetics of the analyzed metals;
* taking medication;
* taking discretionary agents (excessive alcohol consumption);
* altered physiological states (pregnancy, strenuous physical exercise, recent meal, stress, psychological disorders);

INCLUSION CRITERIA:

* age: subjects of working age, between 28 and 70 years;
* diagnosis of Parkinson's disease (using the criteria of the "London Brain Bank")

Ages: 28 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases: subjects of both sexes with at least 10 years of work seniority with diagnosis of Parkinson's disease, coming from Neuromed IRCCS and Second University of Naples Controls: healthy subjects matched by age, sex, lifestyle habits and areas of residence, work seniority.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Enrollment | two-year
  Enrollment: In order to verify if some factors might be connected with a metals exposure for the disease onset, a questionnaire investigating the patients' residence area, the field of work and the specific activities carried out, as well as lifestyle habits has been prepared.
  Sample Collection: Patients and controls will be subject to blood sampling for manganese, copper and iron quantitative analysis
Sample Collection | two-year
  We sample 5 ml of blood in tube serum (at least 2 ml of serum) then we label the test tube with an identifying code which is: S-PRK(for cases affected by Parkinson followed by a progressive number es. S-PRK 1,2,3…..), and S-CRL (for controls followed by a progressive number es. S-CRL 1,2,3….)
  This samples will be centrifugated at 4000 rpm for 10 min. Than we divide the serum in 5 eppendorf of 1.5 mL for cases and 5 for controls:
  * Eppendorf 1: 300 µl of serum labeled AMN-X (X indicating the progressive number both for cases and controls)
  * Eppendorf 2: 300 µl of serum labeled BMN-X
  * Eppendorf 3: 300 µl of serum labeled ACU-X
  * Eppendorf 4: 300 µl of serum labeled BCU-X
  * Eppendorf 5: the remaining serum put in Fe-X
  The aliquots will be stored in a refrigerator at 4-6 ° C (no longer than 7 days) in appropriate Eppendorf box, in order to avoid the inclination of the sample with consequent loss of serum.

SECONDARY OUTCOMES:
determination by atomic absorption spectroscopy of the concentration of manganese, copper and iron | two-year
  the determination by atomic absorption spectroscopy of the concentration of manganese, copper and iron on the eppendorf sampled will be carried out at the Laboratory of Industrial Toxicology of Occupational Medicine Area - Section of Hygiene, Occupational Medicine, Forensic Medicine of the Second University of Naples

OTHER OUTCOMES:
The statistical data analysis using the SPSS software | two-year
  Statistical analysis will be carry out by using the SPSS software, version 14.0.1 for Windows (SPSS ITALIA s.r.l Bologna, Italy)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Pedata, researcher, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (2):
- Italy (2):
  - Neuromed IRCCS, Pozzilli, Isernia
  - Second University of Naples, Naples, Napoli